CLINICAL TRIAL: NCT01121939
Title: Phase II Study of the Combination of Bevacizumab, Pertuzumab, and Sandostatin for Patients With Advanced Neuroendocrine Cancers.
Brief Title: Combination of Bevacizumab, Pertuzumab, and Sandostatin for Adv. Neuroendocrine Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 135
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2015-09-23 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Neuroendocrine Carcinoma
Keywords: advanced neuroendocrine; Gastrointestinal; Bevacizumab; Avastin; Pertuzumab; Omnitarg; 2C4; Sandostatin; Octreotide
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Bevacizumab; pertuzumab; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): combination of bevacizumab, pertuzumab, and sandostatin for patients with advanced neuroendocrine cancers
  Interventions: Drug: Bevacizumab; Drug: Pertuzumab; Drug: Sandostatin LAR® Depot

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg IV Day 1. The first dose should be administered over
  90 minutes. If no adverse reactions occur after the initial dose, the second dose should
  be administered over a minimum of 60 minutes. If no adverse reactions occur after the
  second dose, all subsequent doses should be administered over a minimum of 30
  minutes. Bevacizumab will be infused prior to pertuzumab.
  Other Names: Avastin
Drug: Pertuzumab — 840 mg IV loading dose infused over 60 minutes. The loading dose is given on Cycle 1, Day 1 or as below. Subsequent doses of pertuzumab are 420 mg IV. If the patient tolerates the initial infusion over 60 minutes, the patient may receive subsequent infusions over 30 minutes. Otherwise, pertuzumab should be infused over 60 minutes. Patients should be observed for 30 minutes after completing the pertuzumab infusion.
  If a patient misses a dose of pertuzumab for 1 cycle (i.e., 2 sequential cycles or administrations are 6 weeks or more apart), a re-loading dose (840 mg) of pertuzumab should be given. If re-loading pertuzumab is administered, subsequent doses of 420 mg will then be given every 3 weeks, starting 3 weeks later.
  Other Names: Omnitarg; 2C4
Drug: Sandostatin LAR® Depot — 30 mg will be given every 28 days by IM injection. The dose of sandostatin may be increased, at the discretion of the treating physician, if necessary to control symptoms related to tumor secretion of vasoactive peptides.
  Other Names: Octreotide

SUMMARY:
The purpose of this Phase II trial will be to define the activity of a VEGF inhibitor

bevacizumab, HER1/HER2 inhibitor pertuzumab, and sandostatin for patients with

advanced neuroendocrine cancers. In particular, the efficacy of bevacizumab and

pertuzumab treatment is of great interest. The primary endpoint of this trial will be

response rate. Toxicity and progression-free survival will be obtained and evaluated.

DETAILED DESCRIPTION:
* To determine overall response rate of patients with low grade neuroendocrine cancer when treated with the combination of bevacizumab, pertuzumab and sandostatin LAR®.
* To determine the disease control rate (objective response + stable disease), time to treatment progression, progression-free survival, and overall survival in patients with advanced low grade neuroendocrine cancer when treated with bevacizumab, pertuzumab and Sandostatin LAR® treatment.
* To define the toxicity and safety of the combination of bevacizumab, pertuzumab and Sandostatin LAR® when used in patients with advanced low grade neuroendocrine cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proven advanced, unresectable or metastatic, well-differentiated (or low-grade) neuroendocrine carcinoma, including typical carcinoid, pancreatic islet cell and other well-differentiated neuroendocrine carcinomas.
2. Patients with documented evidence of disease progression.
3. Patients currently receiving or previously treated with single agent Sandostatin LAR® are eligible.
4. Patients must have >=1 unidimensional measurable lesion definable by

   MRI or CT scan. Disease must be measurable per RECIST version 1.1 criteria.
5. Left Ventricular Ejection Fraction (LVEF) >=50% as determined by either ECHO or MUGA <=6 weeks prior to study entry.
6. An ECOG Performance Status of 0-2.
7. Laboratory values as follows:

   * ANC >=1500/μL
   * Hgb >=9 g/dL
   * Platelets >=100,000/μL
   * AST/SGOT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases
   * ALT/SGPT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases
   * Bilirubin <=1.5 x ULN
   * Creatinine <=2.0 mg/dL or calculated creatinine clearance >=50 mL/min
8. Patients >=18 years of age.
9. Patients must have a life expectancy >12 weeks.
10. Patient must be accessible for treatment and follow-up.
11. Women of childbearing potential must have a negative serum or urine pregnancy test performed <=7 days prior to start of treatment. Women of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
12. Patients must be able to understand the nature of the study and give

written informed consent, and comply with study requirements

Exclusion Criteria:

1. Patients with poorly differentiated neuroendocrine carcinoma, highgrade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid, atypical carcinoid, anaplastic carcinoid, and small cell carcinoma are not eligible.
2. Previous treatment with VEGF or EGFR inhibitors.
3. Cytotoxic chemotherapy, immunotherapy or radiotherapy <=4 weeks prior to study entry.
4. History or known presence of central nervous system (CNS) metastases.
5. Patients who have had a major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury <=4 weeks prior to beginning treatment.
6. Female patients who are pregnant or lactating.
7. History of hypersensitivity to active or inactive excipients of any component of treatment (bevacizumab, sandostatin, and/or pertuzumab).
8. Patients with proteinuria at screening as demonstrated by urine dipstick for proteinuria >=2+ (patients discovered to have >=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection, and must demonstrate <=1 g of protein/24 hours to be eligible).
9. Patients with a serious non-healing wound, active ulcer, or untreated bone fracture.
10. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
11. Patients with history of hematemesis or hemoptysis (defined as having bright red blood of ½ teaspoon or more per episode) <=1 month prior to study enrollment.
12. History of myocardial infarction or unstable angina <=6 months prior to beginning treatment.
13. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and /or diastolic blood pressure >100 mmHg while on antihypertensive medications). Initiation of antihypertensive agents is permitted provided adequate control is documented at least 1 week prior to Day of study treatment.
14. New York Heart Association (NYHA) grade II or greater congestive

    heart failure (CHF).
15. Serious cardiac arrhythmia requiring medication.
16. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) <=6 months prior to Day 1 of treatment.
17. History of stroke or transient ischemic attack <=6 months prior to beginning treatment.
18. Any prior history of hypertensive crisis or hypertensive encephalopathy.
19. History of abdominal fistula or gastrointestinal perforation <=6 months prior to Day 1 of beginning treatment.
20. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
21. Any known positive test for human immunodeficiency virus, hepatitis C virus or acute or chronic hepatitis B infection.
22. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
23. Use of any non-approved or investigational agent <=28 days prior to administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
24. Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS >=5 years.
25. Infection requiring IV antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, S.B., M.D., Study Chair — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Baptist Medical Center East, Louisville, Kentucky
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Tennessee Oncology Associates, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Bevacizumab: 15 mg/kg IV Day 1. The first dose should be administered over
  90 minutes. If no adverse reactions occur after the initial dose, the second dose should
  be administered over a minimum of 60 minutes. If no adverse reactions occur after the
  second dose, all subsequent doses should be administered over a minimum of 30
  minutes. Bevacizumab will be infused prior to pertuzumab.
  Pertuzumab: 840 mg IV loading dose infused over 60 minutes. The loading dose is given on Cycle 1, Day 1 or as below. Subsequent doses of pertuzumab are 420 mg IV. If the patient tolerates the initial infusion over 60 minutes, the patient may receive subsequent infusions over 30 minutes.
  Sandostatin LAR® Depot: 30 mg will be given every 28 days by IM injection.
Period: Overall Study
Arm/Group | All Patients
Started | 43
Completed | 0 (Patients remained on-study until disease progression or unacceptable toxicity occurred.)
Not Completed | 43

BASELINE CHARACTERISTICS:
Population: All Patients
Arm/Group | All Patients
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: Includes all patients
Measure: Number; unit: percentage of participants
Groups:
- Typical Carcinoid: Patients with typical carcinoid disease
- Pancreatic Islet Cell: Patients with pancreatic islet cell disease
- All Patients: All patients on study (treatment is same for all patients)
Arm/Group | Typical Carcinoid | Pancreatic Islet Cell | All Patients
Number analyzed (Participants) | 32 | 11 | 43
percentage of participants | 16 | 18 | 16

2. Secondary Outcome: Define Toxicity and Safety
Description: To define the toxicity and safety of the combination of bevacizumab, pertuzumab and Sandostatin LAR® when used in patients with advanced low grade neuroendocrine cancer - defined by grade 3/4, treatment-related toxicity
Time Frame: 18 months
Population: All patients on study
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 43
participants
  Hypertension | 11
  Pain | 5
  Left ventricular systolic dysfunction | 5
  Diarrhea | 3
  Anemia | 1
  Leukopenia | 1

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Population: Includes all patients (patients in both the typical carcinoid and pancreatic islet cell groups received the same treatment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Typical Carcinoid | Pancreatic Islet Cell
Number analyzed (Participants) | 32 | 11
months | 11.96 [3.9 to 15.7] | 5.49 [1.1 to 6.5]

4. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Typical Carcinoid | Pancreatic Islet Cell
Number analyzed (Participants) | 32 | 11
months | NA [22.4 to NA] — Median OS and upper bound of 95% confidence interval not reached (NR) at this time | 26.4 [3.0 to NA] — Upper bound of 95% confidence interval not reached (NR) at this time

5. Secondary Outcome: Disease Control Rate
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment or Experience Stable Disease. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither Sufficient Shrinkage to Qualify For PR, Nor Sufficient Increase to Qualify for Progressive Disease; Disease Control Rate = CR + PR + SD.
Time Frame: 18 months
Population: Includes all patients
Measure: Number; unit: percentage of participants
Arm/Group | Typical Carcinoid | Pancreatic Islet Cell | All Patients
Number analyzed (Participants) | 32 | 11 | 43
percentage of participants | 72 | 91 | 77

ADVERSE EVENTS:
Time Frame: 18 months
Description: Includes adverse events of all grades, regardless of their relationship to study treatment
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 6/43
Other Adverse Events (participants affected / at risk) | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=43)
Abdominal Pain (Gastrointestinal disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Colonic Obstruction (Gastrointestinal disorders) | 1
Creatinine Increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Kidney Infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 2
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) - Other, Carcinoid Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=43)
Diarrhea (Gastrointestinal disorders) | 27
Fatigue (General disorders) | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18
Headache (Nervous system disorders) | 18
Hypertension (Vascular disorders) | 18
Nausea (Gastrointestinal disorders) | 17
Proteinuria (Renal and urinary disorders) | 16
Anemia (Blood and lymphatic system disorders) | 13
Vomiting (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 9
Abdominal Pain (Gastrointestinal disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 8
Aspartate Aminotransferase Increased (Investigations) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 7
Mucositis (Gastrointestinal disorders) | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Edema Limbs (General disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Weight Loss (Investigations) | 6
Alkaline Phosphatase Increased (Investigations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Creatinine Increased (Investigations) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Insomnia (Psychiatric disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5
Platelet Count Decreased (Investigations) | 5
Sinusitis (Infections and infestations) | 5
Alanine Aminotransferase Increased (Investigations) | 4
Bloating (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Ejection Fraction Decreased (Investigations) | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Musculoskeletal And Connective Tissue Disorders - Other, Body Ache (Musculoskeletal and connective tissue disorders) | 4
Rash Acneiform (Skin and subcutaneous tissue disorders) | 4
White Blood Cell Decreased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Blood Bilirubin Increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Fever (General disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 3
Flushing (Vascular disorders) | 3
Gastrointestinal Disorders - Other, Stomatitis (Gastrointestinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Infections And Infestations - Other, Unknown (Infections and infestations) | 3
Injury, Poisoning And Procedural Complications - Other, Abrasion (Injury, poisoning and procedural complications) | 3
Investigations - Other, Blood Urea Nitrogen Increased (Investigations) | 3
Pain (General disorders) | 3
Rectal Hemorrhage (Gastrointestinal disorders) | 3
Rectal Pain (Gastrointestinal disorders) | 3
Skin Infection (Infections and infestations) | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3
Upper Respiratory Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 3
Watering Eyes (Eye disorders) | 3
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Anxiety (Psychiatric disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 2
Depression (Psychiatric disorders) | 2
Edema (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Heart Failure (Cardiac disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Hot Flashes (Vascular disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Injection Site Reaction (General disorders) | 2
Investigations - Other, Blood Protein Decreased (Investigations) | 2
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 2
Nail Infection (Infections and infestations) | 2
Oral Hemorrhage (Gastrointestinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 2
Respiratory, Thoracic And Mediastinal Disorders - Other, Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, Thoracic And Mediastinal Disorders - Other, Runny Nose (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis Infective (Infections and infestations) | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other, Cold Sores (Skin and subcutaneous tissue disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other, Nail Changes (Skin and subcutaneous tissue disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Wound Complication (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites